CLINICAL TRIAL: NCT00540241
Title: Performance Status and Influencing Factors During Second-Line Treatment With Pemetrexed in Patients With Stage III/IVNon Small Cell Lung Cancer
Brief Title: Performance Status During Treatment With Pemetrexed in Patients With NSCLC
Acronym: PERFORMANCE
Status: Completed | Type: Observational
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Other Study IDs: 11826; H3E-SB-B007 (Other: Eli Lilly and Company)
Record Dates: First submitted 2007-10-04; First posted 2007-10-05 (Estimated); Last update posted 2011-03-29 (Estimated); Status verified 2011-03

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Second-line pemetrexed treatment in NSCLC: Patients with NSCLC who will start second-line treatment with pemetrexed.
  Interventions: Drug: Pemetrexed

INTERVENTIONS:
Drug: Pemetrexed — in-label use
  Other Names: Alimta

SUMMARY:
The primary research objective of this observational study in pretreated patients with NSCLC of Stage IIIa/b or Stage IV is to evaluate patients' Karnofsky Index (KI) after the second cycle of second-line treatment with single agent pemetrexed in a real life setting, and to evaluate factors potentially influencing performance status in terms of KI, i.e. frequency of use of concomitant medications, in particular analgesics, folic acid, Vitamin B12, antiemetics, and medications against diarrhea; as documented in patient diary (days of use per week) and by the physicians.

ELIGIBILITY:
Inclusion Criteria:

* Are 18 years of age or older
* Have NSCLC, Stage IIIa/b or IV, that is not amenable to curative therapy
* Have had one prior chemotherapy regimen with cytotoxic agents for the treatment of NSCLC (patients with adjuvant and neoadjuvant regimens are also eligible. However, patients with one prior cytotoxic chemotherapy followed by a targeted agent such as erlotinib are not eligible because the targeted agent would be regarded as second-line treatment)
* Are initiating second-line of treatment for NSCLC with pemetrexed
* Have been fully informed and have given written consent for the use of their data.

Exclusion Criteria:

* Have received any prior treatment with pemetrexed
* Are participating in a study including administration of any investigational drug or procedure at entry into this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with NSCLC Stage IIIa/b or IV who have previously been treated with chemotherapy and are starting second-line treatment with single-agent pemetrexed are eligible for this observational study. Patients must have received one prior chemotherapy regimen. Patients who received prior neoadjuvant or adjuvant therapy are also eligible. Both, in- and outpatients are eligible.
Sampling Method: Non-Probability Sample
Enrollment: 542 (Actual)
Dates: Start 2007-09; Primary Completion 2009-10 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bad Homburg, Germany

REFERENCES:
- [Derived] Schuette W, Tesch H, Buttner H, Krause T, Soldatenkova V, Stoffregen C. Second-line treatment of stage III/IV non-small-cell lung cancer (NSCLC) with pemetrexed in routine clinical practice: evaluation of performance status and health-related quality of life. BMC Cancer. 2012 Jan 13;12:14. doi: 10.1186/1471-2407-12-14. PMID 22244076
- See also: (Lilly Clinical Trial Registry) — http://lillytrials.com